CLINICAL TRIAL: NCT03898700
Title: Coaching in Context for Caregivers of Children With Spinal Cord Injury
Brief Title: Coaching for Caregivers of Children With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 533863
Record Dates: First submitted 2019-01-22; First posted 2019-04-02 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Pre-post coaching intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- coaching in context (Other): 10, 1 hour sessions of face to face strength based coaching sessions provided face to face or over the phone.
  Interventions: Behavioral: strength based coaching

INTERVENTIONS:
Behavioral: strength based coaching — strength based and solution focused coaching

SUMMARY:
This pilot study has two aims. The first aim is to establish the feasibility of coaching for caregivers of youth with spinal cord injury, and the second aim is to establish methodological procedures for a future multi-center study on the effectiveness of coaching as an intervention for caregivers of youth with spinal cord injury.

DETAILED DESCRIPTION:
This study addresses the unmet needs of female primary informal caregivers of youth with spinal cord injury. A one-group pre-post treatment design will be used. Consented caregivers will receive coaching via face-to-face or via the phone. Each caregiver will participate in up to 10 coaching sessions. Each coaching session will last up to 90 minutes. Coaching sessions will be audiorecorded and transcribed verbatim. Outcomes of coaching on caregivers' self-identified goals will be assessed using the Canadian Occupational Performance Measure.

ELIGIBILITY:
Inclusion Criteria:

* female primary caregiver of youth between 6-13 years of age with traumatic spinal cord injury
* female primary caregivers have legal guardianship of their child with spinal cord injury
* speak, read and comprehend English
* be available for face-to-face coaching
* have a cell phone with text messaging capabilities, and willing to utilize cell or land line for coaching and data collection
* able to verbalize changes in their own participation or their child's participation during initial screen
* written consent

Exclusion Criteria:

* severe mental health condition of female caregiver, as documented in child's medical record or reported to research staff by child's treating MD or medical team member
* abuses illicit or prescribed substances or alcohol at time of initial screen as documented in child's medical record or reported to research staff by child's treating MD or medical team member

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study is focused on primary female informal caregivers
Enrollment: 9 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MJ Mulcahey, PhD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - Shriners Hospitals for Children, Chicago, Illinois
  - Shriners Hospitals for Children, Philadelphia, Pennsylvania
  - TIRR Memorial Hermann Rehabilitation Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Coaching in Context: 10, 1 hour sessions of strength based coaching sessions provided face to face or via phone
  strength based coaching: strength based and solution focused coaching
Period: Overall Study
Arm/Group | Coaching in Context
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Coaching in Context: 10, 1 hour sessions of strength based coaching sessions
  strength based coaching: strength based and solution focused coaching
Arm/Group | Coaching in Context
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.14 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Canadian Occupational Performance Measure [Mean (Full Range); unit: units on a scale] — Semi-structure interview in which clients identified goals for coaching. For each goal, performance and satisfaction are scored on a scale between 1-10, where 1 is "cannot do" and "very unsatisfied" and 10 is "can do without a problem" and "very satisfied". The mean performance and satisfaction scores for each participant are calculated, and the mean of the means is calculated for group scores.
  units on a scale
    Performance Score | 4.23 [1 to 8]
    Satisfaction Score | 3.97 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Canadian Occupational Performance Measure (COPM)
Description: Rates self perceived performance and satisfaction with self-identified goals on a 10 point likert scale (1 cannot do, not satisfied; 10 can do without a problem, very satisfied). A 2-point change is considered clinically meaningful.
Time Frame: Baseline - before coaching and repeated at end of 10 coaching sessions (12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coaching in Context
Number analyzed (Participants) | 7
score on a scale
  COPM Performance | 2.48 (2.01)
  COPM Satisfaction | 2.80 (1.33)
Statistical Analysis 1: Comparison: Coaching in Context; This one-group feasibility study examined outcomes of coaching using descriptive statistics (changed score) and the Wilcoxon signed-rank test. A changed score of 2 points reflects clinical significance. The Wilcoxon was used to determine statistical significance. Performance scores from 31 coaching goals across 7 informal caregivers were used for analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2
Statistical Analysis 2: Comparison: Coaching in Context; This one-group feasibility study examined outcomes of coaching using descriptive statistics (changed score) and the Wilcoxon signed-rank test. A changed score of 2 points reflects clinical significance. The Wilcoxon was used to determine statistical significance. Satisfaction scores from 31 coaching goals across 7 informal caregivers were used for analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 2

ADVERSE EVENTS:
Time Frame: up to 10 weeks
Description: 10 Coaching sessions were provided over a period of up to 10 weeks, during which time adverse events were monitored.
Groups:
- Coaching in Context: 10, 1 hour sessions of strength based coaching via phone.
  strength based coaching: strength based and solution focused coaching
Arm/Group | Coaching in Context
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
We did not achieve our desired sample size of 16. We originally planned to have an equal number of caregivers in each group, however caregivers did not want to be coached in person due to logistical challenges. The study is limited by the small sample size, and COPM scores were generated from more than one goal from each caregiver (there were 31 COPM goals across the 7 participants, with each participant contributing between 3-5 goals).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT03898700/Prot_SAP_000.pdf